CLINICAL TRIAL: NCT05625399
Title: A Phase 3, Randomized, Open-label, Study of Subcutaneous Nivolumab + Relatlimab Fixed-dose Combination Versus Intravenous Nivolumab + Relatlimab Fixed-dose Combination in Participants With Previously Untreated Metastatic or Unresectable Melanoma
Brief Title: A Study of Subcutaneous Nivolumab + Relatlimab Fixed-dose Combination (FDC) in Previously Untreated Metastatic or Unresectable Melanoma
Acronym: RELATIVITY-127
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA224-127; 2022-000575-39 (EudraCT Number); U1111-1274-0193 (Registry Identifier: WHO)
Record Dates: First submitted 2022-11-15; First posted 2022-11-22 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Melanoma
Keywords: Nivolumab; Relatlimab; FDC; Melanoma; rHuPH20; OPDUALAG
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; relatlimab; Opdualag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab + Relatlimab FDC SC (Experimental)
  Interventions: Drug: Nivolumab + Relatlimab; Drug: rHuPH20
- Nivolumab + Relatlimab FDC IV (Active Comparator)
  Interventions: Drug: Nivolumab + Relatlimab

INTERVENTIONS:
Drug: Nivolumab + Relatlimab — Specified dose on specified days
  Other Names: BMS-986213; Opdualag
Drug: rHuPH20 — Specified dose on specified days
  Arms: Nivolumab + Relatlimab FDC SC

SUMMARY:
The purpose of this study is to demonstrate that the study drug exposure level of the nivolumab + relatlimab FDC subcutaneous (SC) formulation is not worse than nivolumab + relatlimab FDC intravenous (IV) administration in participants with previously untreated metastatic or unresectable melanoma.

ELIGIBILITY:
Inclusion Criteria

* Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1/Lansky Performance Score ≥ 80% for adolescents (≥ 12 to < 18 years of age).
* Participants must have histologically confirmed Stage III (unresectable) or Stage IV (metastatic) melanoma, per the American Joint Committee for Cancer (AJCC) staging system.
* Participants must have measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
* Participants must be ≥ 12 years of age. Participants who are ≥ 12 years of age and < 18 years of age (adolescents) must weigh ≥ 40 kg at the time of signing the informed consent (assent).
* Participants must have histologically confirmed Stage III (unresectable) or Stage IV (metastatic) melanoma, per the AJCC staging system (8th edition).

Exclusion Criteria

* Participants must not have ocular melanoma.
* Participants must not have a history of myocarditis, regardless of etiology.
* Participants must not have a condition requiring systemic treatment with either corticosteroids (>10 milligrams [mg] daily prednisone equivalent) or other immunosuppressive medications within 14 days of start of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses >10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 579 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2027-11-18 (Estimated)

PRIMARY OUTCOMES:
Time-averaged serum concentration over 28 days after the first dose (Cavgd28) of Nivolumab | Up to 28 days
Trough serum concentration at steady state (Cminss) of Nivolumab | Up to 4 months
Cavgd28 of Relatlimab | Up to 28 days
Cminss of Relatlimab | Up to 4 months

SECONDARY OUTCOMES:
Objective Response Rate (ORR) by Blinded Independent Central Review (BICR) per RECIST v1.1 | Up to approximately 3 years
Trough serum concentration at Day 28 after the first dose (Cmind28) of Nivolumab and Relatlimab | Up to 28 days
Peak serum concentration after the first dose (Cmax1) of Nivolumab and Relatlimab | Up to 28 days
Time to Cmax1 (Tmax1) of Nivolumab and Relatlimab | Up to 28 days
Peak serum concentration at steady state (Cmaxss) of Nivolumab and Relatlimab | Up to 4 months
Time-averaged serum concentration at steady state (Cavgss) of Nivolumab and Relatlimab | Up to 4 months
Duration of Response (DOR) by BICR per RECIST v1.1 | Up to approximately 3 years
Disease Control Rate (DCR) by BICR per RECIST v1.1 | Up to approximately 3 years
Time to Response (TTR), by BICR per RECIST v1.1 | Up to approximately 3 years
Objective Response Rate (ORR) by Investigator per RECIST v1.1 | Up to approximately 3 years
DOR by Investigator per RECIST v1.1 | Up to approximately 3 years
DCR by Investigator per RECIST v1.1 | Up to approximately 3 years
TTR by Investigator per RECIST v1.1 | Up to approximately 3 years
Progression Free Survival (PFS) by BICR and Investigator per RECIST v1.1 | Up to approximately 3 years
Overall Survival | Up to approximately 3 years
Number of Participants with Adverse Events (AEs) | Up to approximately 3 years
Change from Baseline in Functional Assessment of Cancer Therapy - Melanoma Subscale (FACT-MS) | Up to approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (149):
- United States (15):
  - Local Institution - 0125, Phoenix, Arizona
  - Local Institution - 0189, Springdale, Arkansas
  - Local Institution - 0098, Los Angeles, California
  - Local Institution - 0093, Orange, California
  - Local Institution - 0123, Stanford, California
  - Local Institution - 0113, Englewood, Colorado
  - Local Institution - 0114, Jacksonville, Florida
  - Local Institution - 0146, Baltimore, Maryland
  - Local Institution - 0071, Rochester, Minnesota
  - Local Institution - 0013, Omaha, Nebraska
  - Local Institution - 0169, Cleveland, Ohio
  - Local Institution - 0139, Easton, Pennsylvania
  - Local Institution - 0124, Philadelphia, Pennsylvania
  - Local Institution - 0122, Murray, Utah
  - Local Institution - 0115, Fairfax, Virginia
- Australia (15):
  - Local Institution - 0050, Coffs Harbour, New South Wales
  - Local Institution - 0175, Orange, New South Wales
  - Local Institution - 0172, Port Macquarie, New South Wales
  - Local Institution - 0118, Wagga Wagga, New South Wales
  - Local Institution - 0184, Waratah, New South Wales
  - Local Institution - 0033, Westmead, New South Wales
  - Local Institution - 0055, Wollstonecraft, New South Wales
  - Local Institution - 0090, Birtinya, Queensland
  - Local Institution - 0008, Bendigo, Victoria
  - Local Institution - 0059, Box Hill, Victoria
  - Local Institution - 0154, Heidelberg, Victoria
  - Local Institution - 0030, Melbourne, Victoria
  - Local Institution - 0109, Traralgon, Victoria
  - Local Institution - 0106, Nedlands, Western Australia
  - Local Institution - 0161, Nedlands, Western Australia
- Austria (4):
  - Local Institution - 0027, Graz
  - Local Institution - 0029, Salzburg
  - Local Institution - 0168, Sankt Pölten
  - Local Institution - 0037, Vienna
- Belgium (3):
  - Local Institution - 0072, Brussels
  - Local Institution - 0078, Charleroi
  - Local Institution - 0016, Liège
- Brazil (12):
  - Local Institution - 0177, Fortaleza, Ceará
  - Local Institution - 0180, Vitória, Espírito Santo
  - Local Institution - 0107, Belo Horizonte, Minas Gerais
  - Local Institution - 0025, Ijuí, Rio Grande do Sul
  - Local Institution - 0031, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0058, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0002, Porto Alegrelegre, Rio Grande do Sul
  - Local Institution - 0159, Blumenau, Santa Catarina
  - Local Institution - 0009, Barretos, São Paulo
  - Local Institution - 0018, São José do Rio Preto, São Paulo
  - Local Institution - 0110, Rio de Janeiro
  - Local Institution - 0130, São Paulo
- Canada (5):
  - Local Institution - 0141, Calgary, Alberta
  - Local Institution - 0121, Hamilton, Ontario
  - Local Institution - 0096, Ottawa, Ontario
  - Local Institution - 0116, Toronto, Ontario
  - Local Institution - 0103, Québec, Quebec
- Chile (9):
  - Local Institution - 0178, Port Montt, Los Lagos Region
  - Local Institution - 0119, Santiago, Providencia
  - Local Institution - 0143, Temuco, Región de la Araucanía
  - Local Institution - 0028, Viña del Mar, Región de Valparaíso
  - Local Institution - 0140, Recoleta, Santiago Metropolitan
  - Local Institution - 0144, Santiago, Santiago Metropolitan
  - Local Institution - 0010, Santiago, Santiago Metropolitan
  - Local Institution - 0074, Santiago, Santiago Metropolitan
  - Local Institution - 0017, Santiago
- Czechia (5):
  - Local Institution - 0083, Prague, NY
  - Local Institution - 0094, Hradec Králové
  - Local Institution - 0091, Olomouc
  - Local Institution - 0082, Ostrava Poruba
  - Local Institution - 0095, Prague
- Finland (3):
  - Local Institution - 0164, Helsinki
  - Local Institution - 0167, Tampere
  - Local Institution - 0162, Turku
- France (15):
  - Local Institution - 0108, Toulouse, Cedex 9
  - Local Institution - 0127, Chambray-lès-Tours, Indre-Et-Loire
  - Local Institution - 0111, Lille, Nord
  - Local Institution - 0063, Nantes, OH
  - Local Institution - 0061, Villejuif, Val-De-Marne
  - Local Institution - 0007, Amiens
  - Local Institution - 0128, Bayonne
  - Local Institution - 0022, Bordeaux
  - Local Institution - 0129, Clermont-Ferrand
  - Local Institution - 0046, Dijon
  - Local Institution - 0117, Marseille
  - Local Institution - 0052, Pierre-Bénite
  - Local Institution - 0089, Rennes
  - Local Institution - 0099, Rouen
  - Local Institution - 0034, Paris, Île-de-France Region
- Germany (19):
  - Local Institution - 0101, Heidelberg, Baden-Wurttemberg
  - Local Institution - 0079, Ulm, Baden-Wurttemberg
  - Local Institution - 0011, Regensburg, Bavaria
  - Local Institution - 0003, Lübeck, Schleswig-Holstein
  - Local Institution - 0060, Berlin
  - Local Institution - 0038, Buxtehude
  - Local Institution - 0136, Dortmund
  - Local Institution - 0039, Erfurt
  - Local Institution - 0049, Essen
  - Local Institution - 0166, Frankfurt am Main
  - Local Institution - 0065, Giessen
  - Local Institution - 0135, Göttingen
  - Local Institution - 0138, Hamburg
  - Local Institution - 0137, Ludwigshafen
  - Local Institution - 0165, Marburg
  - Local Institution - 0044, Minden
  - Local Institution - 0112, Nuremberg
  - Local Institution - 0053, Rostock
  - Local Institution - 0081, Tübingen
- Israel (5):
  - Local Institution - 0026, Afula
  - Local Institution - 0054, Jerusalem
  - Local Institution - 0102, Petah-Tikvah
  - Local Institution - 0173, Tel Aviv
  - Local Institution - 0035, Tel Litwinsky
- Italy (7):
  - Local Institution - 0051, Bari
  - Local Institution - 0077, Genova
  - Local Institution - 0170, Milan
  - Local Institution - 0084, Napoli
  - Local Institution - 0032, Perugia
  - Local Institution - 0064, Roma
  - Local Institution - 0014, Siena
- Norway (4):
  - Local Institution - 0163, Bodø
  - Local Institution - 0156, Grålum
  - Local Institution - 0158, Lørenskog
  - Local Institution - 0155, Oslo
- Poland (5):
  - Local Institution - 0171, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Local Institution - 0021, Krakow, Lesser Poland Voivodeship
  - Local Institution - 0005, Opole, Opole Voivodeship
  - Local Institution - 0015, Poznan, Wiekopolskie
  - Local Institution - 0066, Warsaw
- Spain (15):
  - Local Institution - 0012, Donostia / San Sebastian, Gipuzkoa
  - Local Institution - 0086, A Coruña
  - Local Institution - 0134, Badalona
  - Local Institution - 0047, Barcelona
  - Local Institution - 0024, Barcelona
  - Local Institution - 0153, Jaén
  - Local Institution - 0045, Las Palmas de Gran Canaria
  - Local Institution - 0040, Madrid
  - Local Institution - 0126, Madrid
  - Local Institution - 0004, Madrid
  - Local Institution - 0056, Madrid
  - Local Institution - 0006, Seville
  - Local Institution - 0041, Valencia
  - Local Institution - 0043, Valencia
  - Local Institution - 0151, Valencia
- Sweden (2):
  - Local Institution - 0062, Solna, Stockholm County
  - Local Institution - 0097, Lund
- Switzerland (3):
  - Local Institution - 0092, Bern
  - Local Institution - 0080, Chur
  - Local Institution - 0105, Lausanne
- United Kingdom (3):
  - Local Institution - 0088, London, Greater London
  - Local Institution - 0068, Headington, Oxford, Oxfordshire
  - Local Institution - 0120, Newcastle upon Tyne, Tyne and Wear

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT05625399.html